CLINICAL TRIAL: NCT07041463
Title: Impact of a New Psychoeducation Program Coordinated by an Advanced Practce Nurse on the Burden of Family Caregivers of Patients With a First Pyschotic Episode.
Brief Title: Psychoeducation Program for Family Caregivers Coordinated by an APRN
Acronym: APIPEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-A00412-47; PHRIP-22-0039 (Other Grant/Funding Number: DGOS FRANCE)
Record Dates: First submitted 2025-05-28; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: First Episode Psychosis (FEP); Caregiver Burden; Nurse Practitioners; IMPACT OF A NEW PSYCHOEDUCATION PROGRAM COORDINATED BY AN ADVANCED PRACTICE NURSE ON THE BURDEN OF FAMILY CAREGIVERS OF PATIENTS WITH A FIRST PSYCHOTIC EPISODE
Keywords: First Episode Psychosis (FEP); Caregiver burden; Advanced Practice Nurse
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled stepped wedge cluster trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation program coordinated by an APRN (Experimental): The intervention includes an APRN reception, listening and orientation consultation, harmonized during a preparatory meeting prior to setting up the study. At the very least, this should include empathetic listening to the young person's problems, a tour of the unit, an explanation of the young person's background and an explanation of the approach.
  * Individual and group psycho-education programs. Each investigating center will be trained in the same tools, in order to harmonize practices:
  * BREF: This is a 3-session psycho-educational program in which each family is received individually by a pair of caregivers who are not involved in the patient's care.
  * PEPs Caregiver: This is a group psycho-education program in 5 2-hour sessions developed in the coordinating center.
  Interventions: Other: Psychoeducation program coordinated by an APRN; Other: Usual Care
- USUAL intervention (Other): The intervention includes an APRN reception, listening and orientation consultation, harmonized during a preparatory meeting prior to setting up the study. At the very least, this should include empathetic listening to the young person's problems, a tour of the unit, an explanation of the young person's background and an explanation of the approach.
  In the control phase, the caregiver will benefit from the interventions and referrals provided for caregivers "as usual" at each center.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Psychoeducation program coordinated by an APRN — Individual and group psycho-education programs. Each investigating center will be trained in the same tools, in order to harmonize practices:
  * BREF: This is a 3-session psycho-educational program in which each family is received individually by a pair of caregivers who are not involved in the patient's care.
  * PEPs Caregiver: This is a group psycho-education program in 5 2-hour sessions developed in the coordinating center.
  Arms: Psychoeducation program coordinated by an APRN
Other: Usual Care — The caregiver will benefit from the interventions and referrals provided for caregivers "as usual" at each center.

SUMMARY:
The aim of this study is to assess the impact of implementing a specific family program coordinated by APRNs, covering the 5 levels of the family care pyramid through a consultation, an individual psychoeducation program and a group psychoeducation program, on improving caregiver burden and thus contributing to the recovery of users suffering from FEP.

Detailed Description: Psychotic disorders are among the most disabling chronic pathologies in psychiatry. These disorders modify the individual's perceptions, thoughts, moods, behaviours and day-to-day functioning (Implementing interventions as early as possible in the first psychotic episode (FEP) would be likely to decrease the severity and consequences of the illness and improve prospects for recovery. Evidence supports the establishment of multidisciplinary teams to detect early and treat early those experiencing FEP and those at increased risk of psychosis. Recommended interventions include cognitive-behavioral therapies, family interventions, employment and educational support, and above all, at the heart of the system, case management. These specialized teams need to be multidisciplinary, bringing together psychiatrists, psychologists and social workers in addition to case managers. More recently in France, Advanced practice nurse (APRN) have joined these teams. But getting young people to accept both disorders and care is a difficult necessity, and remains a major challenge. Poor compliance with treatment is said to be one of the primary causes of relapse after FEP. Factors that increase the risk of relapse include initially more severe symptoms, persistent substance abuse, poor adherence to treatment and inadequate support from family and friends. Nowadays, support from a close caregiver for a person living with a psychic disorder is recognized as a very favorable factor for long-term prognosis. But the occurrence of a FEP often has the effect of a tidal wave for loved ones, who present high levels of psychological distress and feelings of burden. Unfortunately, it is still difficult for families to gain access to family caregiver support services, which are still insufficiently available and often unknown to them. A number of barriers stand in the way of systematically proposing family interventions, such as health professionals' lack of awareness of the effectiveness of interventions aimed at family carers, their difficulty in establishing a double therapeutic alliance with the young person and his or her family, or the misperception that family interventions are in contradiction with professional secrecy.

The pyramid of family care in early intervention presents the family support that should be available to families of young people with FEP. The levels of intervention are designed to meet the support needs of family caregivers and can be used flexibly depending on specific needs or the phase of the psychotic episode. Also, APRNs could contribute to the success of these caregiver support programs thanks to their skills in prevention, assessment and coordination of complex pathways. This study therefore aims to determine the extent to which a specific program coordinated by APRNs can influence the burden of a family caregiver of a young person suffering from FEP.

DETAILED DESCRIPTION:
Implementing a specific family program coordinated by APRNs, covering the 5 levels of the family care pyramid through a consultation, an individual psychoeducation program and a group psychoeducation program, on improving caregiver burden and thus contributing to the recovery of users suffering from FEP.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver relative of a patient under the care of the FEP team and meeting the criteria of international recommendations of FEP diagnosis made by the specialized team of less than 6 months, between 18 and 35 years of age.
* Caregiver having received information about the study and having giveń consent.
* Caregiver covered by a health insurance plan

Exclusion Criteria:

* Caregiver under curatorship, guardianship, safeguard of justice, family habilitation or future protection mandate
* Caregiver participating in another study that may interact with this one
* Caregiver not fluent in French (comprehension/reading)
* Caregiver who has already received psycho-education on FEP
* Patient's opposition to caregiver's participation in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2029-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Caregiver's burden | 2 times : Baseline and at 6 months
  The ZARIT scale is a validated, self-reported questionnaire that assesses the emotional, physical and financial burden of caring for a sick person. It consists of 22 items, with response modalities on a Likert scale), rated from 0 to 4, giving a score from 0 to 88. A low score represents a limited level of perceived burden, while a high score reflects a heavy burden.

SECONDARY OUTCOMES:
Caregiver's burden | 2 times : at 3 months and at 12 months
  Change in ZARIT score of caregiver between inclusion and 3 months, between inclusion and 12 months the same as primary outcome measure
The mood of the caregiver | 4 times : at inclusion, at 3 months, at 6 months and at 12 months
  The CES-D (center of epidemiologic studies depression) scale is a self-administered questionnaire that assesses the subject's mood by asking how often, in the past week, he or she has experienced symptoms or behaviors associated with depression. Symptom frequency is measured using a 4-point Likert scale (0=never to 3=frequently). The overall score ranges from 0 to 60. Higher scores correspond to more severe symptoms
The caregiver's personal effectiveness | 4 times : at inclusion, at 3 months, at 6 months and at 12 months
  General Self-Efficacy Scale GSE French version. This is a self-administered questionnaire where each statement refers to a successful adaptation and implies a stable internal attribution of success. It uses a 1-4 response scale of "Not at all true" "Barely true", "Moderately true" and "Totally true". The total score is calculated by adding up the responses to each statement: it can therefore vary from 10 to 40.
Quality of life for caregivers | 2 times : at inclusion, at 12 months
  The World Health Organization Quality of Life WHOQOL-BREF. This 26-item questionnaire is completed by the respondent. It comprises 4 domains: "physical health", "psychological well-being", "social relationships" and "environment". Items are answered using a five-level scale (from "not at all" to "rather no", 'about', "most of the time" to "completely"). The scales are highly internally consistent.
Involvement in patient care | 2 times : at inclusion, at 12 months
  The Service Engagement Scale SES. This is a 14-point measure that assesses service-user engagement from the staff's point of view. The case manager involved in the service user's care assesses his or her agreement with the statements using a four-point Likert scale about the user's availability, collaboration with the user, help-seeking and adherence to treatment.
User recovery | 2 times : at inclusion, at 12 months
  The Stages Of Recovery Instrument STORI. This self-administered questionnaire assesses the stage of recovery reached by a patient with a psychotic disorder. The STORI is made up of 50 items, presented in 10 groups of 5. Each group represents one of the four recovery processes (Hope, Identity, Meaning, Responsibility).
Implementation of the intervention | 1 time : at 12 months
  Acceptability: rate of acceptance of participation in the study by family caregivers, number of refusals and early stops in the program, proportion of family caregivers benefiting from the entire program
Acceptance of study participation | 1 time : at 12 months
  Acceptance of study participation by caregivers will be measured by the proportion of caregivers who agreed to participate in the study among those who were offered the study
Feasibility of the program | 1 time at 12 months
  Feasibility of the program will be measured by the average length of time between stages of the program
qualitative evaluation of the implementation | 1 time : at 12 months
  qualitative evaluation of the implementation during semi-structured interviews with the APRNs at each center and the family caregivers in the experimental group. This qualitative survey will enable us to determine satisfaction with the program, understand the perceived effects of the program and its acceptability, and explore the perceived obstacles and limitations of the program and its implementation. These elements will be studied at both individual (caregivers, users and professionals) and organizational (services, environment) levels. The posture, missions and role of the APRNs with patients, families and within the FEP team will be studied in semi-directed interviews.
Program transferability | 1 time : at 12 months
  Program transferability (the extent to which the effects of an intervention in one context can be observed in another) will be analyzed using the Tool for Analyzing Transferability and Supporting the Adaptation of Health Promotion InteRventions (ASTAIRE Grid). This tool assesses the transferability of an intervention based on the characteristics of the target population, the environment in which the intervention is implemented and the support required for transfer
The relapse | 1 time : at 12 months
  Relapse will be defined as any general worsening of the person's condition (decline in level of functioning) requiring intervention such as hospitalization, day hospital follow-up or mobile team intervention for the duration of study participation
Adherence to the program | 1 time : at 12 months
  Adherence to the program will be measured by the percentage of participants who completed the program among all caregivers included.
The fidelity of the program | 1 time at 12 months
  The fidelity of the program delivered will be measured by the number of sessions of the program delivered compared with the initial program.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHRU de Brest - Hôpital de BOHARS,, Bohars
  - CH le Vinatier, Bron
  - Groupe Hospitalier Marius Lacroix, La Rochelle
  - Hôpital La Colombière, Montpellier
  - CHU de Nîmes, Nîmes